CLINICAL TRIAL: NCT07329348
Title: Comparison of Accentuated Eccentric and Concentric Resistance Training on Aerobic Capacity and Strength in Athletes.
Brief Title: Comparison of Accentuated Eccentric and Concentric Resistance Training in Athletes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0481
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Sports Physical Therapy
Keywords: Accentuated Eccentric; concentric; resistance training

STUDY DESIGN:
Intervention Model Description: randomized cinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The AERT group performed eccentric resistance training by Elastic Resistance bands for 3 sessions per week for 8 weeks. Each session included 3 sets of 10 repetitions with 2-3 mints of rest interval between each set. Participants in this group start with Yellow band (light resistance) and progressing through to purple band (high resistance). The level of exercise progressively increased throughout the 8-week program, by increasing the resistance of resistance bands. In group A, participants executed the Eccentric Phase for 2-4 seconds and Concentric phase for 1-2 seconds.
  Interventions: Other: Accentuated eccentric resistance training ( group A)
- Group B (Experimental): The CRT group performed concentric resistance training by Elastic Resistance bands for 3 sessions per week for 8 weeks. Each session included 3 sets of 10 repetitions with 2-3 mints of rest interval between each set. Participants in this group start with Yellow band (light resistance) and progressing through to purple band (high resistance). The level of exercise progressively increased throughout the 8-week program, by increasing the resistance of resistance bands. In group B, participants executed the Concentric Phase for 2-4 seconds and Eccentric phase for 1-2 seconds.
  Interventions: Other: Concentric Resistance training (group B)

INTERVENTIONS:
Other: Accentuated eccentric resistance training ( group A) — The AERT group performed eccentric resistance training by Elastic Resistance bands for 3 sessions per week for 8 weeks. Each session included 3 sets of 10 repetitions with 2-3 mints of rest interval between each set. Participants in this group start with Yellow band (light resistance) and progressing through to purple band (heavy resistance). The level of exercise progressively increased throughout the 8-week program, by increasing the strength of resistance bands. In group A, participants executed the Eccentric Phase for 2-4 seconds and Concentric phase for 1-2 seconds. 12 Comparison of accentuated eccentric and concentric resistance training in athletes
  Arms: Group A
Other: Concentric Resistance training (group B) — The CRT group performed concentric resistance training by Elastic Resistance bands for 3 sessions per week for 8 weeks. Each session included 3 sets of 10 repetitions with 2-3 mints of rest interval between each set. Participants in this group start with Yellow band (light resistance) and progressing through to purple band (heavy resistance). The level of exercise progressively increased throughout the 8-week program, by increasing the strength of resistance bands. In group B, participants executed the Concentric Phase for 2 4 seconds and Eccentric phase for 1-2 seconds.
  Arms: Group B

SUMMARY:
This study will be randomized clinical trial and will recruit male soccer players aged 18-30yrs.Participants will be randomly divided into two groups with each group performing their program 3 times per week for 8 weeks.Group A will engage in Accentuated Eccentric resistance training ,using resistance bands and Group B will participate in Concentric Reistance training ,with similar resistance bands.

DETAILED DESCRIPTION:
Study Design: Randomized Clinical Trials Sample size: 78(39 for each group) Sampling technique: Non-probability, Purposive sampling technique

Study Setting:

* Pakistan Football Federation, Lahore
* Model town soccer club, Lahore

Inclusion criteria:

* Male soccer players
* Age 18 to 30 years.
* A minimum of two years of experience in Regular training
* Athletes with BMI 18.5kg/m2 -24.9kg/m2

Exclusion criteria:

* History of lower extremity surgeries (e.g., ACL reconstruction or any major surgery) in the past year
* Athletes having consumption of Drugs which may influence Athlete performance.
* Any systemic illness
* Any musculoskeletal disorder
* Pre-existing Cardiovascular and respiratory (exercise-induced asthma) conditions

Tools:

* Aerobic capacity:20-meter shuttle run test (ICC =0.96)
* Muscle strength :1RM Back squat test (ICC=0.91-0.99)

ELIGIBILITY:
Inclusion Criteria:

* • Male soccer players

  * Age 18 to 30 years.
  * A minimum of two years of experience in Regular training
  * Athletes with BMI 18.5kg/m2 -24.9kg/m2

Exclusion Criteria:

* • History of lower extremity surgeries (e.g., ACL reconstruction or any major surgery) in the past year

  * Athletes having consumption of Drugs which may influence Athlete performance.
  * Any systemic illness
  * Any musculoskeletal disorder
  * Pre-existing Cardiovascular and respiratory (exercise-induced asthma) conditions

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
1-RM Back Squat test | 8 weeks
  a warm up of 10 repetitions using an empty barbell in back squat position. After rest of 2 mints, Participants will perform same protocol with addition of (35 pounds) weight and goal is to perform maximum repetitions. At final phase, weight (35 pounds) and the maximum repetitions performed are counted. This count is then used in Epley formula to calculate the individual 1RM (32).
  Epley's Formula:
  1RM = weight x (1 + (reps / 30))
20-MTR Shuttle Run test | 8 weeks
  The 20-meter shuttle run test, often called the "beep" or "bleep" test, requires participants to run back and forth continuously between two lines 20 meters apart, with a rhythm imposed by audio(beep). Starting at a slow pace, they must turn when signaled by the beeps. After about a minute, the pace increased, with the beeps occurring more quickly, requiring the runners to speed up. The speed increases each minute(level), with beeps becoming closer together. If a participant reaches the line before the beep, they must wait; if not, they receive a warning and have two more chances to catch up to the pace. A second warning results in elimination from the test. Calculation: VO2max = 18.043461 + (0.3689295 x TS) + (- 0.000349 x TS x TS)

CONTACTS AND LOCATIONS:
Overall Officials: ayesha aslam, DPT, Principal Investigator — Riphah International University; Muhammad faheem Afzal, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Model Town Football Club, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Teoldo I, Dambroz F, Brito J. Performance of soccer players under acute physical fatigue: An approach based on cognitive, tactical and physical aspects. Heliyon. 2024 Apr 30;10(9):e30516. doi: 10.1016/j.heliyon.2024.e30516. eCollection 2024 May 15. PMID 38726114
- [Background] Businari GB, de Camargo JBB, Barbosa PH, Brigatto FA, Aoki MS, Braz TV, Lopes CR. Chronic Effects of Heavy Load Activity Performed Before Resistance Training Sessions on the Physical Performance of Youth Soccer Players. Int J Exerc Sci. 2022 Feb 1;14(6):1421-1434. doi: 10.70252/SDEL8387. eCollection 2021. PMID 35514743
- [Background] Leao C, Silva AF, Badicu G, Clemente FM, Carvutto R, Greco G, Cataldi S, Fischetti F. Body Composition Interactions with Physical Fitness: A Cross-Sectional Study in Youth Soccer Players. Int J Environ Res Public Health. 2022 Mar 18;19(6):3598. doi: 10.3390/ijerph19063598. PMID 35329288
- [Background] Almaawi A, Awwad W, Bamugaddam A, Alasheikh M, Muaddi M, Almutair O, Alomar AZ. Prevalence of knee injuries among male college students in Riyadh, Kingdom of Saudi Arabia. J Orthop Surg Res. 2020 Mar 31;15(1):126. doi: 10.1186/s13018-020-01638-1. PMID 32238180
- [Background] Tayfur B, Charuphongsa C, Morrissey D, Miller SC. Neuromuscular Function of the Knee Joint Following Knee Injuries: Does It Ever Get Back to Normal? A Systematic Review with Meta-Analyses. Sports Med. 2021 Feb;51(2):321-338. doi: 10.1007/s40279-020-01386-6. PMID 33247378